CLINICAL TRIAL: NCT00926575
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Safety and Efficacy of orBec® (Oral Beclomethasone 17,21-Dipropionate)in Conjunction With Ten Days of High-Dose Prednisone Therapy in the Treatment of Patients With Gastrointestinal GVHD
Brief Title: Study of orBec® With Prednisone Therapy in the Treatment of Patients With Graft Versus Host Disease (GVHD)
Acronym: SUPPORTS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: An independent Data Safety Monitoring Board recommended the study be stopped due to futility
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDP-GVHD-03
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-08

CONDITIONS: Acute Gastrointestinal Graft vs Host Disease
Keywords: BDP; orBec; GVHD; beclomethasone dipropionate; bone marrow transplant; hematopoietic cell transplant; HCT; stem cell transplant; marrow transplant; SCT; beclomethasone 17,21-dipropionate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- orBec® (Experimental): Investigational drug
  Interventions: Drug: oral beclomethasone 17,21-dipropionate
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral beclomethasone 17,21-dipropionate — Two tablets QID for 50 days
  Other Names: orBec; BDP
  Arms: orBec®
Drug: Placebo — Two tablets QID for 50 days
  Arms: Placebo

SUMMARY:
Use of an oral topically-active glucocorticoid with limited side effects will control the gastrointestinal inflammatory process of GVHD and minimize glucocorticoid exposure.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of allogeneic hematopoietic cell transplant
* Diagnosis of GI graft vs. host disease (GVHD)
* No GI infection
* Must be able to swallow tablets
* Must be able to read and understand informed consent
* Adequate birth control methods for the duration of the study

Exclusion Criteria:

* Significant Skin GVHD
* Liver GVHD
* Persistent vomiting
* HIV positive
* Pregnancy/lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sullivan, MD, Principal Investigator — Duke University; David Hockenbery, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (3):
- United States (3):
  - Buffalo, New York
  - Durham, North Carolina
  - Seattle, Washington

REFERENCES:
- [Background] McDonald GB, Bouvier M, Hockenbery DM, Stern JM, Gooley T, Farrand A, Murakami C, Levine DS. Oral beclomethasone dipropionate for treatment of intestinal graft-versus-host disease: a randomized, controlled trial. Gastroenterology. 1998 Jul;115(1):28-35. doi: 10.1016/s0016-5085(98)70361-0. PMID 9649455
- [Background] Hockenbery DM, Cruickshank S, Rodell TC, Gooley T, Schuening F, Rowley S, David D, Brunvand M, Berryman B, Abhyankar S, Bouvier M, McDonald GB. A randomized, placebo-controlled trial of oral beclomethasone dipropionate as a prednisone-sparing therapy for gastrointestinal graft-versus-host disease. Blood. 2007 May 15;109(10):4557-63. doi: 10.1182/blood-2006-05-021139. Epub 2007 Jan 23. PMID 17244684

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: oral beclomethasone 17,21-dipropionate (BDP)
Period: Overall Study
Arm/Group | Active | Placebo
Started | 70 | 70
Completed | 54 | 53
Not Completed | 16 | 17
Not completed — Adverse Event | 1 | 1
Not completed — Death | 4 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 8 | 9

BASELINE CHARACTERISTICS:
Population: DSMB terminated study for futility; no safety concerns during analysis of patient population. Overall, 1 SAE considered possibly related to study drug, all others were not related to study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 66 | 128
  >=65 years | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 70
  Male | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With GVHD Treatment Failure
Description: The primary endpoint is the occurrence (yes, no) during the 80-day study period of GVHD treatment failure defined as use of prednisone or equivalent IV corticosteroids at doses higher than stated in the protocol, or use of any additional other glucocorticoid (including unblinded BDP) or addition of other immunosuppressant medications, in response to uncontrolled signs or symptoms of GVHD
Time Frame: Day 80
Population: Data was not analyzed as the study was terminated due to futility
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cumulative Exposure to Prednisone
Time Frame: Day 80
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Survival Status
Time Frame: Day 200
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 80
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 32/70 | 28/70
Other Adverse Events (participants affected / at risk) | 70/70 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=70) | Placebo (N=70)
Acute myeloid leukemia progression (Blood and lymphatic system disorders) | 0 | 1
Angiopathic Anemia (Blood and lymphatic system disorders) | 0 | 1
Leukemic Relapse (Blood and lymphatic system disorders) | 0 | 1
Multiple myeloma progression (Blood and lymphatic system disorders) | 1 | 0
Recurrent AML (Blood and lymphatic system disorders) | 1 | 0
Relapsed ALL (Blood and lymphatic system disorders) | 0 | 1
Relapsed AML (Blood and lymphatic system disorders) | 0 | 1
Thrombotic Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Diabetic Ketoacidosis (Endocrine disorders) | 1 | 0
Disease Progression (General disorders) | 1 | 1
Drug Withdrawal Syndrome (General disorders) | 0 | 1
DVT (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 2 | 1
Flank Pain (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Progressive disease (General disorders) | 0 | 1
Abdominal Cramps (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Increased Abdominal Cramping (Gastrointestinal disorders) | 0 | 1
Intermittent Diarrhea (Gastrointestinal disorders) | 0 | 1
Intractable Nausea (Gastrointestinal disorders) | 0 | 1
Intractable vomiting (Gastrointestinal disorders) | 0 | 1
Loose Stool (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Peritoneal Perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Watery Diarrhea (Gastrointestinal disorders) | 1 | 0
Acute GVHD flare (Immune system disorders) | 1 | 0
Lower GI GVHD (Immune system disorders) | 0 | 1
Back Pain (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
BK Viruria (Infections and infestations) | 1 | 0
BK Virus Cystitis (Infections and infestations) | 0 | 1
BK Virus Infection (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
CMV infection (Infections and infestations) | 2 | 0
CMV infection/reactivation (Infections and infestations) | 1 | 0
CMV Pneumonitis (Infections and infestations) | 1 | 0
CMV reaction (Infections and infestations) | 1 | 0
CMV Reactivation (Infections and infestations) | 0 | 1
Gram Negative Bacilli Hyperbilirubinemia (Infections and infestations) | 1 | 0
Gram Negative Bacteremia (Infections and infestations) | 1 | 0
Gram Positive Bacteremia (Infections and infestations) | 1 | 0
Lower Extremities Cellulitis (Infections and infestations) | 0 | 1
Nocardia sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Right orbital cellulitis (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic Pneumonia (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Skin GVHD (Infections and infestations) | 1 | 0
Staph Bacteremia (Infections and infestations) | 1 | 0
Viral Respiratory-type Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
RSV Positive (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Poor PO Intake (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain: Bone Diffuse (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Meningismus (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Acute Renal Failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Acute Respiratory Distress with Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachyarrhythmia absoluta (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension Worsened (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.43% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=70) | Placebo (N=70)
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 7 | 7
Trombocytopenia (Blood and lymphatic system disorders) | 9 | 6
Tachycardia (Cardiac disorders) | 4 | 6
Adrenal insufficiency (Endocrine disorders) | 4 | 3
Dry Eye (Eye disorders) | 7 | 1
Vision Blurred (Eye disorders) | 5 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 20 | 14
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 33 | 17
Dry Mouth (Gastrointestinal disorders) | 9 | 8
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Flatulence (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 22 | 21
Retching (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 12 | 17
Asthenia (General disorders) | 7 | 6
Early Satiety (General disorders) | 4 | 1
Chills (General disorders) | 2 | 3
Fatigue (General disorders) | 17 | 22
Oedema (General disorders) | 3 | 2
Oedema Peripheral (General disorders) | 6 | 8
Pyrexia (Gastrointestinal disorders) | 12 | 9
Acute graft versus host disease in skin (Immune system disorders) | 5 | 5
Hypogammagluobulinaemia (Immune system disorders) | 6 | 3
Bacteraemia (Infections and infestations) | 6 | 1
BK virus infection (Infections and infestations) | 5 | 2
Clostridial infection (Infections and infestations) | 4 | 0
Cytomegalovirus infection (Infections and infestations) | 15 | 11
Cytomegalovirus viraemia (Infections and infestations) | 5 | 4
Epstein- Barr virus infection (Infections and infestations) | 4 | 1
Staphylococcal infection (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Blood Creatinine increased (Investigations) | 5 | 5
Breath sounds abnormal (Investigations) | 3 | 1
Hepatic enzyme increased (Investigations) | 3 | 0
Blood lactate dehyrogenase increase (Investigations) | 1 | 3
Neutrophil count increased (Investigations) | 0 | 3
Protein total decreased (Investigations) | 1 | 3
Transaminases increased (Investigations) | 2 | 4
Weight decreased (Investigations) | 8 | 5
Anorexia (Metabolism and nutrition disorders) | 7 | 3
Cushingoid (Metabolism and nutrition disorders) | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 16 | 13
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Fluid retension (Metabolism and nutrition disorders) | 3 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 9 | 9
Neuropathy peripheral (Nervous system disorders) | 2 | 4
Tremor (Nervous system disorders) | 7 | 8
Anxiety (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 9 | 9
Dysuria (Renal and urinary disorders) | 3 | 5
Haematuria (Renal and urinary disorders) | 3 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 1
Renal failure (Renal and urinary disorders) | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epstaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 9 | 10
Rash Macular (Skin and subcutaneous tissue disorders) | 2 | 3
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 19 | 7
Hypotension (Vascular disorders) | 3 | 4

LIMITATIONS AND CAVEATS:
DSMB terminated study for futility; no safety concerns during analysis of patient population. Overall, 1 SAE considered possibly related to study drug, all others were not related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other